CLINICAL TRIAL: NCT00038051
Title: Phase I Evaluation of the Anti-CD-33 Immunotoxin Hum-195/rGel in Patients With Advanced Myeloid Malignancies
Brief Title: Evaluation of the Anti-CD-33 Immunotoxin Hum-195/rGel in Patients With Advanced Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-342
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myeloproliferative Disorders; Anemia, Refractory, With Excess of Blasts
Keywords: Acute Myeloid Leukemia; AML; Chronic Myelomonocytic Leukemia; CMML; Myeloproliferative Disorders; Refractory Anemia with Excess of Blasts; RAEB-t; RAEB; Hum-195/rGel
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Anemia, Refractory, with Excess of Blasts | interventions — HuM195-gelonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuM195/rGel (Experimental): HuM195/rGel starting Dose = 3 mg/m^2 twice weekly for 2 weeks.
  Interventions: Drug: Hum-195/rGel

INTERVENTIONS:
Drug: Hum-195/rGel — Starting Dose = 3 mg/m^2 twice weekly for 2 weeks.

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the anti-CD33 immunotoxin HuM-195/rGel that can be given to patients with advanced myeloid malignancies. This treatment will be given to patients whose leukemia has not responded to prior chemotherapy.

DETAILED DESCRIPTION:
Before therapy, all patients will be asked about their medical history, and a physical exam (with measurement of vital signs) will be performed. A chest X-ray and an electrocardiogram (ECG - a test to measure the electrical activity of the heart) will be performed. Blood (about 4 teaspoons) will be drawn for routine tests and blood clotting tests. Women who are able to become pregnant will have a urine pregnancy test done. A test will be done to measure the amount of oxygen in your blood by placing a monitoring device on your finger. Blood (about 1 teaspoon) will be taken to measure the amount of a protein that is present on the diseased cells. During the study period, the study staff will draw blood samples for routine tests, pharmacokinetic (PK) tests, and anti-drug antibody tests. Blood (about 1 teaspoon) will be drawn to measure the amount of a protein that is present on the diseased cells. A bone marrow sample will also be obtained before treatment and on Study Day 28.

Patients will receive four injections of the immunotoxin. The immunotoxin is designed to selectively destroy myeloid leukemia cells. The injections will be given through a vein twice weekly for two weeks. Patients will then be evaluated twice weekly for the next two weeks. If there has been improvement in the leukemia, or if the leukemia has remained stable and there have been no serious side effects of treatment, patients will then receive a second course of immunotoxin injections. These will again be given twice weekly for two weeks. Depending on the effectiveness against leukemia and the side effects, patients may receive maintenance treatment. This would also consist of two weekly injections given for two weeks followed by two weeks of observation. Maintenance therapy may continue for up to four months for partial response and up to two months for complete response.

This is an investigational study. Up to 36 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory acute myelogenous leukemia (AML), Refractory anemia with excess blasts in transformation (RAEB-t), Refractory Anemia with Excess Blasts (RAEB), or chronic myelomonocytic leukaemia (CMML) who failed at least one previous chemotherapy course. Patients with accelerated CML Ph+ or myeloid blastic crisis are eligible. Patients in accelerated phase of non-Philadelphia chromosome + myeloproliferative disorders are also eligible:

   * P. vera,
   * myelofibrosis
   * essential thrombocytopenia with >5% blasts in the blood or bone marrow.
2. Male or female 18 yrs of age or older who have provided written informed consent
3. Tumor cells must be = or > 80% CD33 positive by flow cytometry
4. For women of childbearing potential (i.e. exclude post-menopausal women, women who have been surgically sterilized), adequate birth control methods must be used. Acceptable birth control methods are limited to oral contraceptives, implants, diaphragm, IUD or spermicide used with a condom
5. White blood count (WBC) count <10,000/ml for AML, MDS, and myeloproliferative disorders and up to 30,000 for accelerated CML
6. No cytotoxic chemotherapy for the two weeks prior to entering the study
7. No evidence of residual toxic effects grade 2 or higher from prior chemotherapy
8. Patients with proven bacterial infection are not eligible until resolution of the infection (patient afebrile, not on steroids). Patients with active fungal infections are eligible only if evidence of response to antifungal medications is documented and they do not have fever exceeding 38°C
9. Creatinine - Patients should have values = or < 1.5 times the upper limit of laboratory normal values
10. Liver function - Patients should have serum bilirubin values = or < 2.0 times the upper limit of laboratory normal values. Patients should have SGOT and/or SGPT levels = or < 2.5 times the upper limit of laboratory normal values
11. Cardiac function - Patients with cardiovascular disease should be < New York Heart Association (NYHA) classification III
12. Pulmonary function - O2 saturation should be = or > 92% without exogenous O2 administered.
13. Neurologic function - Patients should have normal central nervous system function as well as normal motor function consistent with = or < Grade 1 toxicity. Patients should have peripheral sensory function damage (neuropathy) not exceeding Grade 1 toxicity

Exclusion Criteria:

Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1999-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Continuous assessment of safety throughout entire study period and determination of dose-limiting toxicities at end of two week evaluation period (4 weeks from start of therapy).
  Dose-limiting toxicity considered to have occurred when (1) >grade 2 extramedullary toxicity possibly related to HuM195/rGel (except nausea, vomiting or diarrhea unless uncontrolled by optimal management, or electrolyte abnormalities unless clinically significant or not correctable after optimal replacement) is observed or (2) >42 days from day 1 of therapy elapse before return of neutrophil count to >500 and platelet count to >25,000 in absence of leukemia (i.e., with a normal or hypercellular bone marrow with <5% blasts).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org